CLINICAL TRIAL: NCT01801007
Title: Pivotal Study of the MicroVention Flow Re-Direction Endoluminal Device (FRED) Stent System in the Treatment of Intracranial Aneurysms
Brief Title: Pivotal Study of the FRED Stent System in the Treatment of Intracranial Aneurysms
Acronym: FRED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL12001; G120111 (Other: FDA)
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-02

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Intervention Model Description: FRED
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flow Re-Direction Endoluminal Device (Other)
  Interventions: Device: Flow Re-Direction Endoluminal Device (FRED)

INTERVENTIONS:
Device: Flow Re-Direction Endoluminal Device (FRED)

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the MicroVention Flow Redirection Intraluminal Device (FRED) system when used in the treatment of wide-necked intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Participant whose age ≥ 22 and ≤75 years
* Participant has single target aneurysm located in the internal carotid artery
* Participant sign and date an IRB/EC approved informed consent prior initiation of any study procedures

Exclusion Criteria:

* Participant who suffers from an intracranial hemorrhage in the last 30 days
* Participant who suffers from a subarachnoid hemorrhage in the last 60 days
* Participant with symptomatic extracranial mass or currently undergoing radiation therapy for tumor of the head and neck region
* Participant who is pregnant or breastfeeding
* Participant has an arteriovenous malformation (AVM) in the area of the target aneurysm

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2013-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cameron McDougall, MD, Principal Investigator — Johns Hopkins University
Locations (24):
- United States (23):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Swedish Medical Center / RIA, Englewood, Colorado
  - Lyerly Neurosurgery, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Norton Neuroscience Institute, Louisville, Kentucky
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Capital Health Hospital, Trenton, New Jersey
  - Albany Medical Center, Albany, New York
  - University at Buffalo, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Health System, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - Baylor Saint Luke Medical Center, Houston, Texas
  - The Methodist Hospital, Houston, Texas
- Institute of Biomedical Research and Innovation, Kobe, Japan

REFERENCES:
- [Derived] McDougall CG, Diaz O, Boulos A, Siddiqui AH, Caplan J, Fifi JT, Turk AS, Kayan Y, Jabbour P, Kim LJ, Hetts SW, Cooke DL, Dowd CF. Safety and efficacy results of the Flow Redirection Endoluminal Device (FRED) stent system in the treatment of intracranial aneurysms: US pivotal trial. J Neurointerv Surg. 2022 Jun;14(6):577-584. doi: 10.1136/neurintsurg-2021-017469. Epub 2021 Jul 19. PMID 34282038

RESULTS

PARTICIPANT FLOW:
Groups:
- Flow Re-Direction Endoluminal Device: The FRED Stent System is intended to be used in the treatment of wide-necked Intracranial Aneurysms.
Period: Overall Study
Arm/Group | Flow Re-Direction Endoluminal Device
Started | 145
Completed | 134
Not Completed | 11
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Flow Re-Direction Endoluminal Device
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 126
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 104
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 139
  Japan | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Occlusion of the Target Aneurysm and ≤50% Stenosis of the Parent Artery and an Alternative Treatment of the Target Intracranial Aneurysm (IA) Had Not Been Performed Within 12 Months
Description: The primary effectiveness endpoint has three components: 1) complete occlusion of the target aneurysm assessed by a core laboratory utilizing the Raymond-Roy Scale 2) ≤ 50% stenosis of the parent artery at the target (IA) using the Warfarin-Aspirin Symptomatic Intracranial Disease(WASID) criterion which is defined as greater than 50% luminal loss, 3) alternative treatment of the target IA is defined as re-treatment of the target aneurysm with an alternative treatment modality including open repair, endovascular placement of an additional stent or treatment of In-stent Stenosis observed. The Raymond-Roy Occlusion Classification has 3 responses, where Grade I is complete occlusion, no flow of contrast seen in the sac, Grade II is partial occlusion, some flow in the neck or sac, and Grade III is incomplete occlusion, apparent flow into the sac. Grade 1 indicates the best outcome.
Time Frame: 12 months
Population: Participants that had 12 month angiographic assessment of vessel stenosis
Measure: Number; unit: percentage of participants
Arm/Group | Flow Re-Direction Endoluminal Device
Number analyzed (Participants) | 139
percentage of participants | 57.0

2. Primary Outcome: Percentage of Participants Who Experience Neurological Death or Major Ipsilateral Stroke Measured by the Modified Rankin Scale (mRS) and the National Institute of Health Stroke Scale (NIHSS)
Description: A major stroke is defined as a new neurological event that persists for > 24 hours and results in a ≥ 4 points increase in the NIHSS score compared to baseline or compared to any subsequent lower score. A major ipsilateral stroke is defined as that occurring within the vascular distribution of the stented artery. Neurologic death is defined as a death which has been adjudicated by the independent clinical events committee to have directly resulted from a neurologic cause.The NIHSS score ranges from 0 (no stroke symptoms) to 42 (severe stroke). mRS is 6 point assessment scale used to assess disability in patients who have suffered a stroke and is compared over time to check for recovery and degree of continued disability. The mRS score ranges from 0 (no disability) to 6 (death).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flow Re-Direction Endoluminal Device
Number analyzed (Participants) | 145
Participants | 9

3. Secondary Outcome: Percentage of Participants With Complete Occlusion of the Target Aneurysm on 12-month Angiography (Raymond-Roy 1)
Description: Complete occlusion of the target aneurysm assessed by a core laboratory. The Raymond-Roy class is an angiographic classification scheme for grading the occlusion (closure) of endovascularly treated intracranial aneurysms: class I: complete obliteration, class II: residual neck, class III: residual aneurysm.
Time Frame: 12 months
Population: Participants that had 12 month angiographic assessment of aneurysm occlusion and vessel stenosis.
Measure: Count of Participants; unit: Participants
Arm/Group | Flow Re-Direction Endoluminal Device
Number analyzed (Participants) | 140
Participants | 88

4. Secondary Outcome: Percentage of Participants With ≥ 50% In-Stent Stenosis (ISS) at the Target Intracranial Aneurysm (IA) at 12 Months as Assessed by Angiography at the Independent Core Laboratory
Description: Stenosis of the parent artery at the target IA using the Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) criterion which is defined as greater than 50% luminal loss
Time Frame: 12 months
Population: Participants that had 12 month angiographic assessment of vessel stenosis.
Measure: Count of Participants; unit: Participants
Arm/Group | Flow Re-Direction Endoluminal Device
Number analyzed (Participants) | 139
Participants | 6

5. Secondary Outcome: Percentage of Participants in Whom an Unplanned Alternative Treatment of the Target IA Had Not Been Performed Within 12 Months
Description: Re-treatment of the target aneurysm with an alternative treatment modality including open repair, endovascular placement of an additional stent or treatment of In-stent Stenosis observed
Time Frame: 12 months
Population: Participants that had 12 months angiographic assessment and vessel stenosis.
Measure: Count of Participants; unit: Participants
Arm/Group | Flow Re-Direction Endoluminal Device
Number analyzed (Participants) | 140
Participants | 132

6. Secondary Outcome: Percentage of Participants With Clinically Acceptable (90-100%) Occlusion of the Target Aneurysm, ≤ 50% Stenosis of the Parent Artery at the Target IA, and an Unplanned Alternative Treatment of the Target IA Had Not Been Performed
Description: This endpoint has three components: 1) clinically acceptable occlusion of the target aneurysm assessed by a core laboratory as percent occlusion (90%-100%) 2) ≤ 50% stenosis of the parent artery at the target IA using the WASID criterion which is defined as greater than 50% luminal loss, 3) alternative treatment of the target IA is defined as re-treatment of the target aneurysm with an alternative treatment modality including open repair, endovascular placement of an additional stent or treatment of In-stent Stenosis observed. The Raymond-Roy scale has 3 responses, where Grade I is complete occlusion, no flow of contrast seen in the sac, Grade II is partial occlusion, some flow in the neck or sac, and Grade III is incomplete occlusion, apparent flow into the sac.
Time Frame: 12 months
Population: Participants that had 12 month angiographic assessment of vessel stenosis.
Measure: Count of Participants; unit: Participants
Arm/Group | Flow Re-Direction Endoluminal Device
Number analyzed (Participants) | 139
Participants | 100

7. Secondary Outcome: Percentage of Participants With Unsuccessful Delivery of the FRED
Description: Inability to deliver a FRED device to the target location
Time Frame: Index Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Flow Re-Direction Endoluminal Device
Number analyzed (Participants) | 145
Participants | 2

8. Secondary Outcome: Percentage of Participants That Had Procedure Related Serious Adverse Events With the FRED System
Description: A serious adverse event is any medical experience regardless of its relationship to the study treatment that occurs during participant enrollment in this trial that results in any of the following: (1) inpatient hospitalization or prolongation of a hospitalization; (b) persistent or significant disability or incapacity; (c) death of the study participant, or (d) necessitates an intervention to prevent a permanent impairment of a body function or permanent damage to a body structure. Procedure related events were associated with the index procedure, antiplatelet therapy, or follow up angiography.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Flow Re-Direction Endoluminal Device
Number analyzed (Participants) | 145
Participants | 40

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Flow Re-Direction Endoluminal Device
All-Cause Mortality (participants affected / at risk) | 2/145
Serious Adverse Events (participants affected / at risk) | 63/145
Other Adverse Events (participants affected / at risk) | 61/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flow Re-Direction Endoluminal Device (N=145)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (3)
Visual impairment (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Device deployment issue (General disorders) | 1 (1)
Device dislocation (General disorders) | 1 (1)
Device failure (General disorders) | 6 (6)
Device malfunction (General disorders) | 1 (1)
Device occlusion (General disorders) | 1 (1)
In-stent cerebral artery stenosis (General disorders) | 1 (1)
Puncture site haemorrhage (General disorders) | 1 (1)
Thrombosis in device (General disorders) | 10 (10)
Abdominal abscess (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Visual field tests abnormal (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Blindness (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 3 (3)
Cerebral hypoperfusion (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 6 (6)
Encephalopathy (Nervous system disorders) | 1 (1)
Eyelid ptosis (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 4 (4)
Mental impairment (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1)
Radiculitis (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 5 (5)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aneurysm repair (Surgical and medical procedures) | 11 (11)
Angioplasty (Surgical and medical procedures) | 1 (1)
Stent placement (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1)
Carotid artery stenosis (Vascular disorders) | 1 (1)
Cerebral vasoconstriction (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Vascular wall hypertrophy (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flow Re-Direction Endoluminal Device (N=145)
Visual impairment (Eye disorders) | 11 (16)
Urinary tract infection (Infections and infestations) | 9 (9)
Headache (Nervous system disorders) | 43 (45)
Haematoma (Vascular disorders) | 9 (9)
Vasospasm (Vascular disorders) | 16 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must inform and submit to sponsor all manuscripts or abstracts at least 30 days prior to submitting the proposed Publication to a publisher or other third party.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT01801007/SAP_000.pdf
  • Study Protocol (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT01801007/Prot_002.pdf